CLINICAL TRIAL: NCT00482742
Title: A Feasibility, Multi Center Multinational Randomized Open Label Study, to Evaluate the Safety and Performance of the CiTop™ Guidewire for Crossing Total Occlusion in Peripheral Arteries.
Brief Title: Safety & Performance Randomized Study of the CiTop™ Guidewire for Peripheral CTO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: product development was cancelled
Sponsor: Ovalum (Industry)
Responsible Party: Principal Investigator, Liat Shochat, investigator, Ovalum
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: OVC-P01-00.CTIL
Record Dates: First submitted 2007-06-03; First posted 2007-06-05 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2013-07

CONDITIONS: Catheterization, Peripheral
Keywords: Chronic Total Occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle counseling (Other)
  Interventions: Device: CiTop(TM) Guidewire
- Metformin (Other)
  Interventions: Device: CiTop(TM) Guidewire

INTERVENTIONS:
Device: CiTop(TM) Guidewire

SUMMARY:
The main objectives of the study are:

To evaluate the performance and safety of the CiTop guidewire, while attempting to cross thru total occlusions of various dimensions and morphology.

To compare the safety and efficacy of the CiTop guidewire with standard guidewires in terms of impact on the treated artery. Following operation of the CiTop device, angiography demonstrated successful crossing of the occlusion with no visible evidence of arterial wall injury, dissection, or distal embolization.

To assess ease of operation and the level of integration of the CiTop with standard interventional angiography procedure: Balloon angioplasty, placement of stent.

ELIGIBILITY:
Clinical Inclusion Criteria:

* Patient with symptomatic peripheral vascular disease, intermittent claudication less than 30 meters, rest pain or tissue ischemia.(Fontain grade 3-4)
* Critical limb Ischemia
* The patient has Chronic Total Occlusion in limb arteries, aged at least 3 months.
* Patient has chronic total occlusion (CTO) that is:
* Documented angiographically, by the investigator or co-investigator.
* CTO was defined as an obstruction of a main peripheral artery with no luminal continuity and with TIMI (Thrombolysis In Myocardial Infraction) flow grade of 0 or 1.
* CTO location suitable for endovascular treatment (not in parallel location with the hip or knee joints).
* Lesion ≤ 8cm in length
* Lesion located in a segment with diameter more than 1.5 mm
* Adequate compliance with follow-up and/or repeat angiography
* No Contra-indication to treatment with aspirin or ticlopidine or clopidogrel and/or Heparin
* Visible entry point of target lesion
* NO cancer or other life threatening diseases or conditions
* NO diagnosis or suspected renal failure (2 x ULN of creatinine)
* Not suspected intolerance of the contrast agent
* NO Drug abuse or alcoholism
* Patients is NOT under custodial care
* Women with childbearing potential are NOT pregnant (positive pregnancy test at the time of procedure).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Belenky, MD, Principal Investigator — Research Fund, Belinson Hospital
Locations (3):
- Croatia (2):
  - University Hospital Split, Split
  - Clinical Hospital Centre Zagreb, Zagreb
- Rabin Campus, Belinson Hospital, Petah Tikva, Israel